CLINICAL TRIAL: NCT01723150
Title: A Multi-centre Randomised Open-label Active Comparator-controlled Non-inferiority Trial Comparing Oral to Intravenous Antibiotics in the Early Management of Klebsiella Pneumoniae Liver Abscess
Brief Title: Antibiotics for Klebsiella Liver Abscess Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Tan Tock Seng Hospital (Other); Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-KLASS
Record Dates: First submitted 2012-10-22; First posted 2012-11-07 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Liver Abscess, Pyogenic
Keywords: Klebsiella pneumoniae
MeSH Terms: conditions — Liver Abscess, Pyogenic | interventions — Ciprofloxacin; Ceftriaxone; Trimethoprim, Sulfamethoxazole Drug Combination; Ertapenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral antibiotics (Experimental): The intervention arm switched to oral antibiotics to complete 4 weeks of therapy. Oral antibiotics will be ciprofloxacin (or trimethoprim/sulfamethoxazole if the isolate is resistant).
  Interventions: Drug: Ciprofloxacin; Drug: Trimethoprim/sulfamethoxazole
- Intravenous antibiotics (Active Comparator): The active comparator arm continues intravenous antibiotics to complete 4 weeks of therapy. Intravenous antibiotics will be ceftriaxone (or ertapenem if the isolate is resistant).
  Interventions: Drug: Ceftriaxone; Drug: Ertapenem

INTERVENTIONS:
Drug: Ciprofloxacin
  Arms: Oral antibiotics
Drug: Ceftriaxone
  Arms: Intravenous antibiotics
Drug: Trimethoprim/sulfamethoxazole
  Other Names: Bactrim
  Arms: Oral antibiotics
Drug: Ertapenem
  Arms: Intravenous antibiotics

SUMMARY:
Background: Klebsiella pneumoniae liver abscess is the most common etiology of liver abscess in Singapore and much of Asia, and its incidence is increasing. Current management includes prolonged intravenous antibiotic therapy, but there is limited evidence to guide oral conversion. The implicated K1/K2 capsule strain of Klebsiella pneumoniae is almost universally susceptible to ciprofloxacin, an antibiotic with high oral bioavailability. Our primary aim is to compare the efficacy of early (<1 week) step-down to oral antibiotics, to continuing 4 weeks of intravenous antibiotics, in patients with Klebsiella liver abscess.

Methods/Design: The study is designed as a multi-centre randomised open-label active comparator-controlled non-inferiority trial, with a non-inferiority margin of 12%. Eligible participants will be inpatients over the age of 21 with a CT or ultrasound scan suggestive of a liver abscess, and Klebsiella pneumoniae isolated from abscess fluid or blood. Randomisation into intervention or active control arms will be performed with a 1:1 allocation ratio. Participants randomised to the active control arm will receive IV ceftriaxone 2 grams daily to complete a total of 4 weeks of IV antibiotics. Participants randomised to the intervention arm will be immediately converted to oral ciprofloxacin 750mg twice daily. At week 4, all participants will have abdominal imaging and be assessed for clinical response (CRP <20 mg/l, absence of fever, plus scan showing that the maximal diameter of the abscess has reduced). If criteria are met, antibiotics are stopped; if not, oral antibiotics are continued, with reassessment for clinical response fortnightly. If criteria for clinical response are met by week 12, the primary endpoint of clinical cure is met. A cost analysis will be performed to assess the cost saving of early conversion to oral antibiotics, and a quality-of-life analysis will be performed to assess if treatment with oral antibiotics is less burdensome than prolonged IV antibiotics.

Discussion: Our results would help inform local and international practice guidelines regarding the optimal antibiotic management of Klebsiella liver abscess. A finding of non-inferiority may translate to the wider adoption of a more cost-effective strategy that reduces hospital length of stay and improves patient-centered outcomes and satisfaction.

ELIGIBILITY:
Inclusion Criteria

1. Inpatient at time of enrollment
2. Age >= 21 years
3. Computed tomography (CT) or ultrasound (US) within the preceding 7 days suggestive of a liver abscess, as defined by presence of one or more focal areas of hypo- or hyper-attenuation within the liver
4. Klebsiella pneumoniae isolated from abscess fluid or blood collected within the preceding 7 days
5. Able and willing to give informed consent

Exclusion Criteria

All subjects meeting any of the following exclusion criteria at baseline will be excluded from participation:

1) Polymicrobial abscess - additional organisms isolated from blood or abscess fluid within the preceding 7 days 2a) Klebsiella pneumoniae resistant to Ceftriaxone AND Ertapenem 2b) Klebsiella pneumoniae resistant to Ciprofloxacin AND Cotrimoxazole 3) On effective* IV antibiotics > 7 days 4a) Hypersensitivity to cephalosporins AND carbapenems; as defined by history of rash, urticaria, angiodema, bronchospasm or circulatory collapse following prior administration.

4b) Hypersensitivity to fluoroquinolones AND sulpha drugs; as defined by history of rash, urticaria, angioedema, bronchospasm or circulatory collapse following prior administration.

4c) History of penicillin anaphylaxis (angioedema, bronchospasm or circulatory collapse). Subjects with a history of only rash or urticaria or unknown reaction to penicillin can be included.

5) Inability to take oral medications for any reason 6) Severe sepsis or septic shock defined as unresolved hypotension (MAP<70) or tachycardia (HR>110), or requirement of inotropic support or ventilation at time of eligibility. Should the subject's hypotension or tachycardia subsequently resolve, and they cease to require inotropes and ventilation within 7 days, they may be reconsidered for eligibility.

7) Established endophthalmitis at time of screening (patients with visual symptoms should have ophthalmology review prior to enrollment) 8) Established central nervous system abscess at time of screening (patients with focal neurology should have CT head prior to enrollment) 9) Women who are pregnant or breastfeeding 10) Inability to obtain consent from subject 11) Patients on tizanidine or theophylline 12) Patients on concomitant drugs that can result in prolongation of the QT interval (e.g., class IA or class III antiarrhythmics) or with risk factors for torsade de pointes (e.g., known QT prolongation, uncorrected hypokalemia) 13) Patients whose K. pneumoniae tests resistant to ciprofloxacin, and those with contraindications to ciprofloxacin will be tested for G6PD deficiency, and excluded if deficient 14) Severe immunocompromise (e.g., active leukemia or lymphoma, generalized malignancy, aplastic anemia, solid organ transplant, bone marrow transplant within 2 years of transplantation, or transplants of longer duration still on immunosuppressive drugs or with graft-versus-host disease, congenital immunodeficiency, current radiation therapy, HIV/AIDS with CD4 lymphocyte count <200 and patients or on immunosuppressant medications) 15) Creatinine clearance <15 ml/min

*defined as antibiotics to which the Klebsiella pneumoniae isolate in blood or abscess fluid is susceptible

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2013-11-05 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2018-01-16 (Actual)

PRIMARY OUTCOMES:
Clinical cure | Week 12
  The primary endpoint is "clinical cure", determined at Week 12 post-randomisation, and defined as CRP< 20 mg/l, plus absence of documented fever ≥38°C in the preceding week, plus most recent abdominal imaging showing that the maximal diameter of the abscess has reduced.

SECONDARY OUTCOMES:
Clinical response | Week 4
  The main secondary endpoint is "clinical response", determined at Week 4 post-randomisation, and defined as CRP <20 mg/l, plus absence of documented fever ≥38°C in the preceding week, plus most recent abdominal imaging showing that the maximal diameter of the abscess has reduced.

OTHER OUTCOMES:
all-cause mortality at any point between randomisation and week 12 | Week 12
• unplanned readmission for any cause at any point between hospital discharge and week 12 | Week 12
• unplanned need for drainage after enrolment at any point between randomisation and week 12 (the screening visit will document any plans for elective drainage) | Week 12
• metastatic complications occurring at any point between randomisation and week 12 | Week 12
new K. pneumoniae bacteraemia occurring at any point between the first negative blood culture, and week 12, with the same strain of K. pneumoniae as the original blood culture or abscess fluid culture | Week 12
• length of hospital stay (from the date of randomisation to the end of inpatient stay, censored at week 12) | Week 12
• length of time the subject requires medical leave following hospital discharge (censored at week 12) | Week 12
• subject quality of life as defined by the WHOQOL-BREF assessed at week 4 and week 12 post-randomisation | Week 12
• overall cost of each treatment strategy from the payer and total societal perspective for the course of the study until the final twelve week follow-up | Week 12
• level of adherence during the entire study period, assessed at twelve weeks. Subject deemed to be compliant if 80% or more of prescribed antibiotics have been taken | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Archuleta, MD, Principal Investigator — National University Hospital, Singapore
Locations (3):
- Singapore (3):
  - Singapore General Hospital, Singapore
  - National University Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore

REFERENCES:
- [Background] Molton J, Phillips R, Gandhi M, Yoong J, Lye D, Tan TT, Fisher D, Archuleta S. Oral versus intravenous antibiotics for patients with Klebsiella pneumoniae liver abscess: study protocol for a randomized controlled trial. Trials. 2013 Oct 31;14:364. doi: 10.1186/1745-6215-14-364. PMID 24176222
- [Derived] Yoong J, Yuen KH, Molton JS, Ding Y, Cher BP, Chan M, Kalimuddin S, Oon J, Young B, Low J, Salada BMA, Lee TH, Wijaya LM, Fisher D, Izharuddin E, Wei Y, Phillips R, Moorakonda R, Lye DC, Archuleta S. Cost-minimization analysis of oral versus intravenous antibiotic treatment for Klebsiella pneumoniae liver abscess. Sci Rep. 2023 Jun 16;13(1):9774. doi: 10.1038/s41598-023-36530-5. PMID 37328522
- [Derived] Molton JS, Chan M, Kalimuddin S, Oon J, Young BE, Low JG, Salada BMA, Lee TH, Wijaya L, Fisher DA, Izharuddin E, Koh TH, Teo JWP, Krishnan PU, Tan BP, Woon WWL, Ding Y, Wei Y, Phillips R, Moorakonda R, Yuen KH, Cher BP, Yoong J, Lye DC, Archuleta S. Oral vs Intravenous Antibiotics for Patients With Klebsiella pneumoniae Liver Abscess: A Randomized, Controlled Noninferiority Study. Clin Infect Dis. 2020 Aug 14;71(4):952-959. doi: 10.1093/cid/ciz881. PMID 31641767